CLINICAL TRIAL: NCT05469893
Title: Immuno-PRISM (PRecision Intervention Smoldering Myeloma): A Randomized Phase II Platform Study of Select Immunotherapies for High-Risk Smoldering Myeloma
Brief Title: Immuno-PRISM (PRecision Intervention Smoldering Myeloma)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Irene Ghobrial, MD (Other)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor-Investigator, Irene Ghobrial, MD, Sponsor Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-154
Record Dates: First submitted 2022-06-07; First posted 2022-07-22 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: High-risk Smoldering Multiple Myeloma; Smoldering Multiple Myeloma; Multiple Myeloma
Keywords: High-risk smoldering Multiple Myeloma; Smoldering Multiple Myeloma; Multiple Myeloma
MeSH Terms: conditions — Smoldering Multiple Myeloma; Multiple Myeloma | interventions — Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lenalidomide + Dexamethasone (LD) (Active Comparator): Each study treatment cycle lasts 28 days. Participants will be randomized into either Teclistamab arm or Lenalidomine + Dexamethoasone arm
  * Lenalidomine
  * Dexamethoasone
  Interventions: Drug: Lenalidomide; Drug: Dexamethasone
- Teclistamab (Experimental): Each study treatment cycle lasts 28 days. Participants will be randomized into either Teclistamab arm or Lenalidomine + Dexamethoasone arm
  - Teclistamab-Per Protocol
  Interventions: Drug: Teclistamab

INTERVENTIONS:
Drug: Teclistamab — Intravenous (IV) dosage and timing per protocol design
  Other Names: JNJ-64007957
  Arms: Teclistamab
Drug: Lenalidomide — Oral, dosage and timing per protocol design
  Other Names: Revlimid
  Arms: Lenalidomide + Dexamethasone (LD)
Drug: Dexamethasone — Oral, dosage and timing per protocol design
  Arms: Lenalidomide + Dexamethasone (LD)

SUMMARY:
The purpose of this study is to test the anti-cancer activity of Teclistamab and to compare it with Lenalidomide + Dexamethasone combination in people with high risk smoldering multiple myeloma.

People with smoldering multiple myeloma (SMM) usually do not have symptoms but are at risk for progressing to active multiple myeloma (MM). Multiple Myeloma is a cancer of the plasma cells, which are an important part of the immune system. Patients with active multiple myeloma generally require treatment but there are currently no approved therapies for smoldering multiple myeloma.

The names of the study drugs involved in this study are:

* Teclistamab
* Lenalidomide (also called Revlimid)
* Dexamethasone (also called Decadron)

DETAILED DESCRIPTION:
This is a multiple arm, randomized, phase II platform study investigating the efficacy of Teclistamab or other immunotherapies against a control arm of Lenalidomide + Dexamethasone combination in participants with high-risk smoldering multiple myeloma.

The names of the study drugs involved in this study are:

* Teclistamab
* Lenalidomide (also called Revlimid)
* Dexamethasone (also called Decadron)

Safety of Teclistamab in SMM population will be established by using safety run-in method in the beginning of the study and will enroll up to 6 participants directly into Teclistamab arm. First 3 participants in cohort 1 will receive lower than recommended phase 2 dose (RP2D) of Teclistamab and will be closely observed for the first 28 days. If safety is established with cohort 1, the additional 3participants will be enrolled to cohort 2 to receive RP2D. Once safety run-in participants indicate that it is safe to proceed, additional participants will be randomized 1:2 to the control arm of Lenalidomide + Dexamethasone combination or an investigational single agent (i.e., Teclistamab) arm. 15 participants will be randomized to the control arm, and 30 participants will be randomized to each investigational drug arm.

This research study has several different stages: screening, treatment, end of treatment and follow up.

The study treatment (either Teclistamab or Lenalidomide + Dexamethasone combination) will continue as long as there is disease benefits from the study drugs or a maximum of 24 months. It is expected that about 51 participants (6 safety + 15 control + 30 investigational arms) will take part in this research study.

Teclistamab and Lenalidomide and Dexamethasone are 'investigational' study drugs, which means that they have not been approved for treatment in high-risk smoldering multiple myeloma in the United States by the Food and Drug Administration (FDA).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* 1) High risk SMM defined as having 1 of the following 2 criteria: High risk per "20-2-20" Criteria defined as presence of any two of the following:

  -- Serum M spike ≥ 2 gm/dL, Involved to uninvolved free light chain (FLC) ratio≥ 20, Bone marrow Plasma Cell (BMPC) % ≥ 20%
* OR total score of 9 using the following scoring system:

  * FLC Ratio >10-25 = 2, >25-40 = 3, > 40 = 5
  * Serum M-Protein (g/dL) >1.5-3 = 3, >3 = 4
  * BMPC% >15-20 = 2, >20-30 = 3, >30-40 = 5, >40 = 6
* Fluorescence In Situ Hybridization (FISH) abnormality (t(4,14), t(14,16), 1q gain, or del13q = 2
* 2) Presence of ≥10% BMPC and at least one of the following:

  -- Evolving pattern:
  * evolving Monoclonal Protein (eMP) (≥10% increase in Monoclonal Protein/Immunoglobulin (Ig)) within the first 6 months (only if M-protein ≥3 g/dl) and/or ≥25% increase in M/Ig within the first 12 months, with a minimum required increase of 0.5 g/dl in M-protein and/or 500 mg/dl in Ig.
  * Evolving change in hemoglobin (eHb) ≥0.5 g/dl decrease within 12 months of diagnosis;
  * Progressive involved light chain increase on two successive evaluation
  * Abnormal Plasma Cell immunophenotype (≥ 95% of BMPCs are clonal) and reduction of ≥1 uninvolved immunoglobulin isotype. (Only IgG; IgA and IgM will be considered)
  * High risk cytogenetics defined as presence of t(4;14), t(14;16), t(14;20), 17p deletion, TP53 mutation, 1q21 gain
  * Monoclonal light chain excretion of > 200mg/24 hours for those with monoclonal light chain SMM
* No evidence of CRAB criteria* or new criteria of active MM (SLIM-CRAB) which include the following:

  * Increased calcium levels: Corrected serum calcium >0.25 mmol/L (>1mg/dL) above the upper limit of normal or >2.75 mmol/L (>11mg/dL);
  * Renal insufficiency (attributable to myeloma);
  * Anemia (Hgb 2g/dL below the lower limit of normal or <10g/dL);
  * Bone lesions (lytic lesions or generalized osteoporosis with compression fractures)
  * No evidence of the following new criteria for active MM including the following:

    * Bone marrow plasma cells >60%
    * Serum involved/uninvolved FLC ratio ≥100
    * MRI with more than one focal lesion
* Participants with CRAB criteria that are attributable to conditions other than the disease under study may be eligible after discussion with the Sponsor Investigator.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0, 1, or 2
* The following laboratory values obtained <28 days prior to registration:

  * Absolute Neutrophil Count (ANC) >1000/mL
  * Platelets Count (PLT) >75,000/mL
  * Total bilirubin ≤ 2.0 mg/dL (If total is elevated check direct and if normal patient is eligible.)
  * Aspartates Aminotransferase (AST) <2.5 x institutional upper limit of normal (ULN)
  * Alanine Transaminase (ALT) <2.5 x institutional upper limit of normal (ULN)
  * Estimated creatinine clearance (CLcr) ≥60 mL/min
* Voluntary written informed consent will be obtained before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Females of child-bearing potential* randomized to Lenalidomide must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days and again within 24 hours prior to prescribing lenalidomide for Cycle 1 (prescriptions must be filled within 7 days as required by Revlimid Risk Evaluation and Mitigation Strategies (REMS®) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide.

  * A female of child-bearing potential is a sexually mature female who: has not undergone a hysterectomy (the surgical removal of the uterus) or bilateral oophorectomy (the surgical removal of both ovaries), or has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time during the preceding 24 consecutive months)
  * A woman must be . A Not of childbearing potential, or b. Of childbearing potential and Practicing true abstinence; or Have a sole partner who is vasectomized; or Practicing ≥1 highly-effective, user-independent method of contraception NOTE: Participant must agree to continue the above throughout the study and for 90 days after the last dose of study treatment.

NOTE: If a woman becomes of childbearing potential after start of the study the woman must comply with point (b) as described above.

NOTE: An interaction between hormonal contraception and teclistamab has not been formally studied. Therefore, it is unknown whether teclistamab may reduce the efficacy of the contraception method.

* A woman must agree not to donate eggs (ova, oocytes) or freeze for future use, for the purposes of assisted reproduction during the study and for 90 days after receiving the last dose of study treatment
* A man must wear a condom (with or without spermicidal foam/gel/film/cream/suppository) when engaging in any activity that allows for passage of ejaculate to another person during the study and for a minimum of 90 days after receiving the last dose of study treatment. If a female partner is of childbearing potential, she must also be practicing a highly effective method of contraception
* If the male participant is vasectomized, he still must wear a condom (with spermicidal foam/gel/film/cream/suppository), but his female partner is not required to use contraception.
* A male participant must agree not to donate sperm for the purpose of reproduction during the study and for a minimum of 90 days after receiving the last dose of study treatment.
* Must be willing and able to adhere to the lifestyle restrictions specified in this protocol
* All study participants randomized to lenalidomide must be registered into the mandatory Revlimid REMS® program and be willing and able to comply with the requirements of the REMS® program.
* Females of child-bearing potential must adhere to the scheduled pregnancy testing as required in the Revlimid REMS® program if randomized to lenalidomide
* Men must agree to use a latex condom during sexual contact with a female of childbearing potential even if they have had a successful vasectomy
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Prior SMM directed therapy administered within 6 months of beginning treatment on study. To avoid including primary refractory cases to the lenalidomide arm, participants who received a prior lenalidomide-based therapy should have had at least an Minimal Response (MR) to be considered on this trial.
* Symptomatic Multiple Myeloma or any evidence of CRAB criteria, including presence of myeloma defining events (MDE). Any prior therapy for active Myeloma should also be excluded. Prior therapy for smoldering myeloma is not an exclusion criterion. Bisphosphonates are not excluded
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational. Prior therapy with bisphosphonate is allowed. Prior radiation therapy to a solitary plasmacytoma is allowed but had to be at least 6 months prior to enrollment on the trial. Prior clinical trials or therapy for smoldering MM or Monoclonal Gammopathy of Unknown Significance (MGUS) are allowed per exclusion criteria described above.
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Diagnosed or treated for another malignancy within 2 years of enrollment
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Plans to father a child while enrolled in this study or within 90 days after receiving the last dose of study drug.
* Pregnant or breast-feeding or planning to become pregnant while enrolled in this study or within 90 days after receiving the last dose of study drug.
* Known seropositive for or active viral infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV) or SARS-CoV-2 (COVID- 19).
* Participants who are seropositive because of hepatitis B virus vaccine are eligible.
* Participants who are positive for SARS-COV-2 antibody, HIV1 and 2 antibody, hepatitis B core antibody or hepatitis B surface antigen must have a negative polymerase chain reaction (PCR) result before enrollment. Those who are PCR positive will be excluded.
* Contraindications or life-threatening allergies, hypersensitivity, or intolerance to any study drug or its excipients (refer to the teclistamab Investigator's Brochure and appropriate package inserts).
* Prior or concurrent exposure to any of the following:
* Investigational vaccine within 4 weeks
* Live, attenuated vaccine within 4 weeks before randomization.
* Monoclonal antibody therapy within 21 days
* Cytotoxic therapy within 14 days
* PI therapy within 14 days
* IMiD agent therapy within 14 days
* Radiotherapy within 14 days or focal radiation within 7 days
* A maximum cumulative dose of corticosteroids of ≥140 mg of prednisone or equivalent within 14-day period before the first dose of study drug (does not include pretreatment medications)
* Known active Central Nervous System (CNS) involvement or exhibits clinical signs of meningeal involvement of multiple myeloma. If either is suspected, negative whole brain MRI and lumbar cytology are required.
* Myelodysplastic syndrome or active malignancies (i.e., progressing or requiring treatment change in the last 24 months). The only allowed exceptions are: a. Non-muscle invasive bladder cancer treated within the last 24 months that is considered completely cured b. Skin cancer (non-melanoma or melanoma) treated within the last 24 months that is considered completely cured. c. Noninvasive cervical cancer treated within the last 24 months that is considered completely cured d. Localized prostate cancer (N0M0): With a Gleason score of ≤6, treated within the last 24 months, or untreated and under surveillance With a Gleason score of 3+4 that has been treated >6 months prior to full study screening and considered to have a very low risk of recurrence, or e. History of localized prostate cancer and receiving androgen deprivation therapy and considered to have a very low risk of recurrence. f. Breast cancer: adequately treated lobular carcinoma in situ or ductal carcinoma in situ, or history of localized breast cancer and receiving antihormonal agents and considered to have a very low risk of recurrence. g. Other malignancy that is considered cured with minimal risk of recurrence
* Stroke or seizure within 6 months prior to signing informed consent form
* Presence of the following cardiac conditions:

  -- New York Heart Association stage III or IV congestive heart failure, 2) Myocardial infarction or coronary artery bypass graft ≤6 months prior to randomization,3) History of clinically significant ventricular arrhythmia or unexplained syncope, not believed to be vasovagal in nature or due to dehydration,4) History of severe non-ischemic cardiomyopathy
* Major surgery within 2 weeks prior to the start of administration of study treatment, or will not have fully recovered from surgery, or has major surgery planned during the time the participant is expected to be treated in the study or within 2 weeks after administration of the last dose of study treatment. NOTE: Participants with planned surgical procedures to be conducted under local anesthesia may participate. Kyphoplasty or vertebroplasty are not considered major surgery. If there is a question whether a procedure is considered a major surgery, the investigator must consult with the appropriate sponsor representative and resolve any issues before enrolling a participant in the study.
* Concurrent medical or psychiatric condition or disease that is likely to interfere with study procedures or results, or that in the opinion of the investigator would constitute a hazard for participating in this study, such as:
* Uncontrolled diabetes defined by Hemoglobin A1C > 8.5, Acute diffuse infiltrative pulmonary disease, Evidence of active systemic viral, fungal, or bacterial infection, requiring systemic, antimicrobial therapy, History of autoimmune disease with the exception of vitiligo, type I diabetes, and, prior autoimmune thyroiditis that is currently euthyroid based on clinical symptoms and laboratory testing, . Disabling psychiatric conditions (e.g., alcohol or drug abuse), severe dementia, or altered mental status, Any other issue that would impair the ability of the participant to receive or tolerate the planned treatment at the investigational site, to understand informed consent or any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (e.g., compromise the wellbeing) or that could prevent, limit, or confound the protocol-specified assessments, History of non-compliance with recommended medical treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2022-08-10 (Actual); Primary Completion 2030-07-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Complete Response Rate (CRR) | Cycle 2 Day 1 through end of follow up (each cycle is 28 days).
  The complete response rate (CRR) was defined as the proportion of participants achieving complete response (CR) based on International Myeloma Working Group (IMWG) Response criteria. CR defined as requires all of the following:
  * Disappearance of the original monoclonal protein from the blood and urine on at least two determinations for a minimum of six weeks by immunofixation studies.
  * <5% plasma cells in the bone marrow on at least two determinations for a minimum of six weeks.
  * No increase in the size or number of lytic bone lesions (development of a compression fracture does not exclude response).
  * Disappearance of soft tissue plasmacytomas for at least six weeks.

SECONDARY OUTCOMES:
Minimal Residual Disease (MRD) Negativity | Baseline, Cycle 6 Day 1, Cycle 13 Day 1, end of treatment, 1, 2, & 3 year after end of treatment (each cycle is 28 day).
  The MRD is expressed as a frequency that quantifies the level of residual disease based on the number of remaining copies of the initially dominant sequence(s) relative to the total number of nucleated cells in the sample.
Progression-free survival (PFS) until progression to myeloma | Every 6 months, up to 3 years after treatment discontinuation.
  Progression-free survival based on the Kaplan-Meier method is defined as the duration of time from study entry to documented disease progression (PD) or death. International Myeloma Working Group (IMWG) Response criteria: Progressive disease (PD) is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. PD for the evaluation of non-target lesions is the appearance of one or more new lesions and/or unequivocal progression of non-target lesions.
Progression-free survival (PFS-2) post initiation of overt myeloma therapy | Every 6 months, up to 3 years after treatment discontinuation.
  Progression-free survivial-2 is defined as time from randomization to disease progression (PD) while receiving overt myeloma therapy, or death from any cause.
Time to progression | Cycle 2 Day1 through end of follow up, an average of 5 years (each cycle is 28 days).
  Time to progression (TTP) is defined as the time of randomization until progression. Participants who have died without evidence of progression are censored in the TTP analysis at the time of death and participants who are alive without progression are censored at the last disease assessment.
Duration of Response (DOR) | Cycle 2 Day1 through end of follow up, an average of 5 years (each cycle is 28 days).
  The duration of overall response is measured as the time from initiation of first response to first documentation of disease progression or death whichever occurs first. Participants who have not progressed or died are censored at the date last known progression-free.
Pharmacodynamic biomarkers of antimyeloma and immune activity of Teclistamab | Cycle 1 Days 1, 8, 9, 11, 15; Cycle 2 Day 1; Cycle 3 & 5 Days 1, 4, 8, and 15; Cycle 12 Day 1; End of treatment; and 8 week after last dose of Teclistamab (each cycle is 28 day).
  Serum from venous blood samples will be collected for measurement of serum concentrations of teclistamab (Arm A - Teclistamab only) and the generation of Anti-drug Antibodies (ADAs) where applicable to teclistamab per the Study Schedule.
Pharmacokinetics of teclistamab in SMM | Cycle 1 Days 1, 8, 9, 11, 15; Cycle 2 Day 1; Cycle 3 & 5 Days 1, 4, 8, and 15; Cycle 12 Day 1; End of treatment; and 8 week after last dose of Teclistamab (each cycle is 28 day).
  Serum from venous blood samples will be collected for measurement of serum concentrations of teclistamab (Arm A - Teclistamab only) and the generation of Anti-drug Antibodies (ADAs) where applicable to teclistamab per the Study Schedule.
Immunogenicity of Teclistamab in SMM | Cycle 1 Days 1, 15; Cycle 3 & 5 Days 1, 4, 8, and 15; and Cycle 12 Day 1 (each cycle is 28 day)
  Serum from venous blood samples will be collected for measurement of serum concentrations of teclistamab (Arm A - Teclistamab only) and the generation of Anti-drug Antibodies (ADAs) where applicable to teclistamab per the Study Schedule.
To assess ability to collect stem cells after Teclistamab | After 4 cycles of treatment; at the time of best response; or at the investigator's discretion as part of standard of care practice.(each cycle is 28 days)
  Stem cell mobilization will be performed with filgrastim alone or filgrastim with plerixafor per institutional standard. In participants that are unable to achieve adequate stem cell yield with filgrastim and plerixafor, cyclophosphamide may be used per institutional standard.
To assess Overall Survival (OS) | Every 6 months up to 3 years after treatment discontinuation.
  OS based on the Kaplan-Meier method is defined as the time from study entry to death or censored at date last known alive.
To assess incidence of Treatment-Emergent Adverse Events that are assessed by the number of patients experiencing at least one treatment-related grade 3 or higher AE of any type during the time of observation | Baseline through end of post-treatment follow up period, an average of 5 years
  All grade 3 or higher adverse events (AE) with treatment attribution of possibly, probably or definite based on Common Terminology Criteria for Adverse Event - Version 5 (CTCAEv5) as reported on case report forms were counted. Incidence is the number of patients experiencing at least one treatment-related grade 3 or higher AE of any type during the time of observation.

CONTACTS AND LOCATIONS:
Overall Officials: Irene C Ghobrial, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Oregon Health & Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu